CLINICAL TRIAL: NCT00005863
Title: Protocol for Patients With High Risk (Resistant, Refractory, Relapsed or Adverse Cytogenetic) AML
Brief Title: Combination Chemotherapy With or Without Filgrastim and/or Tretinoin in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067895; MRC-LEUK-AML-HR; EU-20008
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2006-01

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; adult acute myeloid leukemia in remission; childhood acute myeloid leukemia in remission; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); childhood acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia with maturation (M2); childhood acute myelomonocytic leukemia (M4); childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); childhood acute erythroleukemia (M6); childhood acute megakaryocytic leukemia (M7); secondary acute myeloid leukemia; de novo myelodysplastic syndromes; adult acute monocytic leukemia (M5b); previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; adult acute minimally differentiated myeloid leukemia (M0); childhood acute minimally differentiated myeloid leukemia (M0); atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Congenital Abnormalities | interventions — Filgrastim; Cytarabine; Daunorubicin; Etoposide; fludarabine phosphate; Tretinoin

INTERVENTIONS:
Biological: filgrastim
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: etoposide
Drug: fludarabine phosphate
Drug: tretinoin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy. It is not yet known whether combination chemotherapy with filgrastim and/or tretinoin is more effective than combination chemotherapy alone for acute myeloid leukemia.

PURPOSE: This randomized phase III trial is studying combination chemotherapy with filgrastim and/or tretinoin to see how well they work compared to combination chemotherapy alone in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare standard induction chemotherapy with cytarabine, daunorubicin, and etoposide vs fludarabine and cytarabine in terms of achievement of remission, reasons for remission failure, duration of remission, survival, toxicity, and supportive care needs in patients with high risk acute myeloid leukemia.
* Determine if the use of filgrastim (G-CSF) or tretinoin administered during and following chemotherapy improves outcome in this patient population.
* Determine the impact of these treatment regimens on quality of life in these patients.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are stratified according to type of disease (resistant vs refractory vs relapsed vs adverse cytogenetic), age (under 15 vs 15 to 29, vs 30 to 49 vs 50-59 vs 60-69 vs 70 and over), performance status, and de novo and secondary leukemia. Patients with relapsed disease are further stratified according to duration of first remission (less than 6 months vs 6 to 12 months vs 12 months and over), and prior transplantation (yes vs no).

Patients are randomized into one of two treatment arms for induction chemotherapy.

* Arm I: Patients receive induction chemotherapy consisting of cytarabine IV every 12 hours on days 1-10, daunorubicin IV on days 1, 3, and 5 and etoposide IV over 1 hour on days 1-5. Patients receive a second course of therapy with cytarabine IV every 12 hours on days 1-8 and daunorubicin and etoposide as in course 1.
* Arm II: Patients receive 2 courses of induction chemotherapy consisting of fludarabine IV over 30 minutes followed by cytarabine IV over 4 hours on days 1-5.

Patients are further randomized into one of two treatment arms for colony stimulating factor therapy.

* Arm I: Patients receive filgrastim (G-CSF) subcutaneously or IV daily beginning on day 1 of each course of induction chemotherapy and continuing until blood counts recover, for up to a maximum of 28 days.
* Arm II: Patients receive no G-CSF during and following induction chemotherapy. Patients are further randomized into one of two treatment arms for retinoid therapy.
* Arm I: Patients receive oral tretinoin daily beginning on day 1 of induction chemotherapy and continuing for up to a maximum of 90 days.
* Arm II: Patients receive no retinoid therapy during and following induction chemotherapy.

Following completion of induction chemotherapy, patients achieving complete remission and blood count recovery may receive subsequent therapy consisting of consolidation chemotherapy and/or autologous or allogeneic transplantation.

Quality of life is assessed at 3 months.

PROJECTED ACCRUAL: Approximately 800-1,000 patients will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML) including de novo or secondary AML, or a preexisting myelodysplastic syndrome

  * Overt resistant disease with more than 15% bone marrow blasts after induction course
  * Primary refractory disease

    * Failure to achieve first complete remission after at least 2 induction courses
  * Relapse from first remission with more than 5% bone marrow blasts
  * Complete or partial remission following 1 induction course with adverse cytogenetic abnormalities at diagnosis
* No acute promyelocytic leukemia
* No chronic myeloid leukemia in blast transformation
* No prior relapse from a second or greater remission

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Creatinine clearance at least 30 mL/min

Other:

* No other active malignancy
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-08; Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D. W. Milligan, MD, Study Chair — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- Birmingham Heartlands Hospital, Birmingham, England, United Kingdom

REFERENCES:
- [Background] Burnett AK, Milligan D, Hills RK, et al.: Does all-transretinoic acid (ATRA) have a role in non-APL acute myeloid leukaemia? Results from 1666 patients in three MRC trials. [Abstract] Blood 104 (11): A-1794, 2004.
- [Result] Milligan DW, Wheatley K, Littlewood T, Craig JI, Burnett AK; NCRI Haematological Oncology Clinical Studies Group. Fludarabine and cytosine are less effective than standard ADE chemotherapy in high-risk acute myeloid leukemia, and addition of G-CSF and ATRA are not beneficial: results of the MRC AML-HR randomized trial. Blood. 2006 Jun 15;107(12):4614-22. doi: 10.1182/blood-2005-10-4202. Epub 2006 Feb 16. PMID 16484584